CLINICAL TRIAL: NCT07286188
Title: Effect of Misoprostol on Fluid Deficit Volume in Hysteroscopic Myomectomy: A Double-Blinded Randomized Controlled Trial
Brief Title: Effect of Misoprostol on Fluid Deficit Volume in Hysteroscopic Myomectomy
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Magdy Milad, MD, Albert B Gerbie Professor, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: #STU00223642
Record Dates: First submitted 2025-12-10; First posted 2025-12-16 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Fibroids, Uterine; Fluid Deficit; Hysteroscopy / Methods
Keywords: fibroids; hysteroscopy; myomectomy; fluid deficit; misoprostol
MeSH Terms: conditions — Leiomyoma; Hypovolemia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Patient, surgeon, and research team are masked.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Misoprostol (treatment aem) (Experimental): Patients will received 800 mcg of misoprostol per rectum prior to procedure.
  Interventions: Drug: Misoprostol Tabets
- Zeebo (Placebo arm) (Placebo Comparator): Patient will receive 4 tablets of placebo (ZEEBO) per rectum prior to procedure.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Misoprostol Tabets — 800 mcg of misoprostol will be administered per rectum to intervention group prior to their scheduled hysteroscopic myomectomy.
  Arms: Misoprostol (treatment aem)
Drug: Placebo — 4 tablets of Zeebo (Microcsrystalline cellulose) placebo tablets will be placed per rectum to prior to undergoing a hysteroscopic myomectomy, for patients assigned to the placebo arm.
  Arms: Zeebo (Placebo arm)

SUMMARY:
The goal of this double blinded randomized control trial is to evaluate the impact of misoprostol on fluid deficit during hysteroscopic myomectomies. The main questions it aims to answer are:

Is there is difference in fluid deficit in patients who receive misoprostol vs placebo pre operatively for hysteroscopic myomectomies?

Participants will be randomized to received 800 mcg of either rectal misoprostol prior to their hysteroscopic myomectomy or 4 tablets of placebo (ZEEBO) prior to their hysteroscopic myomectomy.

DETAILED DESCRIPTION:
Misoprostol is a synthetic analogue of prostaglandin E1 originally developed for the prevention and treatment of NSAID-induced peptic ulcers. Over time, it has become widely used in obstetrics and gynecology due to its uterotonic properties. It is FDA-approved as part of the regimen, paired with mifepristone, for medical abortion and is commonly used off-label for cervical ripening, management of postpartum hemorrhage, and preoperative preparation for gynecologic procedures. In non-pregnant women, misoprostol is frequently administered prior to procedures such as hysteroscopy, intrauterine device insertion, and endometrial biopsy to facilitate cervical dilation. It can be delivered via multiple routes, including oral, sublingual, buccal, vaginal, and rectal. Rectal administration typically results in onset of action within 10-20 minutes, peak plasma concentrations at 60-80 minutes, and a duration of action of approximately 3-4 hours due to its short half-life (20-40 minutes). Its uterotonic effects are mediated by increased intracellular calcium, which activates myosin light-chain kinase. Reported side effects include cramping, bleeding, fever, shivering, nausea, vomiting, and diarrhea, though these are generally mild and dose dependent. Previous studies have evaluated misoprostol's ability to reduce intraoperative blood loss during abdominal and laparoscopic myomectomy, typically using a single preoperative administered vaginally or rectally. These studies demonstrated significant reductions in blood loss. In gynecologic practice, doses ranging from 400 to 1000 mcg are commonly used and well tolerated.

Our study focuses on hysteroscopic myomectomy, a minimally invasive procedure performed via the cervix using a hysteroscope to visualize and resect submucosal fibroids within the uterine cavity. Unlike abdominal or laparoscopic approaches, hysteroscopic procedures are not associated with significant blood loss. Instead, the primary intraoperative concern is fluid overload. This can occur when the distension medium, typically normal saline (NS), is absorbed systemically through exposed vascular channels. Although NS is isotonic and does not disrupt electrolyte balance, excessive absorption can lead to complications such as pulmonary edema, cardiac strain, and peripheral edema. To mitigate this risk, national and institutional guidelines recommend terminating the procedure when the fluid deficit (the difference between the volume instilled and the volume recovered) reaches 2.5 liters.

Misoprostol's uterotonic properties may help reduce fluid absorption by promoting uterine contractions and limiting vascular exposure, potentially allowing the procedure to be more complete without exceeding fluid safety thresholds. This potential benefit is biologically plausible and clinically relevant. We have selected a dose of 800 mcg rectally, which is within the established safe and commonly used range in gynecologic practice. This dose is expected to be well tolerated and does not increase risk to participants.To maintain blinding, participants in the placebo arm will receive four Zeebo-branded tablets, each containing 250 milligrams, in weight, of microcrystalline cellulose, administered rectally to match the appearance and administration of the active drug. Zeebo is an inert placebo with no pharmacologic activity, and additional risks are minor.

STUDY ENDPOINTS:

Primary endpoint:

• Difference in intraoperative fluid deficit (in milliliters) as measured by the automated fluid management system, between the misoprostol and placebo groups.

Secondary endpoints:

* Difference in total fluid volume used (in milliliters) between groups.
* Difference in total procedure time (in minutes) between groups.
* Frequency of repeat hysteroscopic myomectomy due to incomplete fibroid resection caused by early termination of the initial procedure.
* Total specimen weight.

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting for hysteroscopic myomectomy for uterine fibroids on pelvic imaging (pelvic ultrasound or MRI) within in last 12 months
* Age ≥ 18 years and ≤ 50 years.
* Fibroids between 1-3cm in size
* Myomectomy using myosure or resectoscope devices
* Willing to have rectal misoprostol or placebo at time of procedure
* Ability to understand and the willingness to sign a written informed consent.
* Admissible medical/surgical history.
* Can be previously treated with Depo-Lupron, Depo-Provera, or Oral Contraceptive pills
* Can have had prior Cesarean delivery

Exclusion Criteria:

* Pregnancy. All patients will be required to have a negative urine pregnancy test prior to surgery.
* Post-menopausal women.
* Patients with a history of gynecologic malignancy.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to misoprostol.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Known active inflammatory bowel disease involving the rectum or other significant anorectal conditions that may interfere with safe rectal administration of study medication.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-12-16 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Fluid Deficit | Immediately at the conclusion of the procedure.
  Primary outcome is difference in fluid deficit at the conclusion of the hysteroscopic myomectomy

SECONDARY OUTCOMES:
Total fluid volume | intraoperative
  Difference in total fluid volume used (in milliliters) between groups.
Time | Intraop
  Difference in total procedure time (in minutes) between groups.
Reoperation | within 3 month post op
  Frequency of repeat hysteroscopic myomectomy due to incomplete fibroid resection caused by early termination of the initial procedure
Specimen weight | Immediately post op
  Total specimen weight

CONTACTS AND LOCATIONS:
Overall Officials: Magy Milad, MD, Principal Investigator — Northwestern University Feinberg School of Medicine, Northwestern Department of Obstetrics and Gynecology, Division of Minimally Invasive Gyn Surgery
Locations (1):
- Northwestern, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No
Plan to present data in aggregate for publication once study completed, individual participant data will not be shared.

REFERENCES:
- [Result] Inacio QAS, Troncon JK, Valerio FP, Herren H, Nogueira AA, Neto OBP, Silva JCRE. Misoprostol Administration Before Hysteroscopy Procedures - A Retrospective Analysis. Rev Bras Ginecol Obstet. 2022 Dec;44(12):1102-1109. doi: 10.1055/s-0042-1755462. Epub 2022 Aug 29. PMID 36037813
- [Result] Guven CM, Avul Z. Evaluation of the effect of preoperative rectal misoprostol use on the postoperative outcomes of hysteroscopic myomectomy. J Obstet Gynaecol Res. 2023 Aug;49(8):2086-2092. doi: 10.1111/jog.15681. Epub 2023 May 19. PMID 37208944
- [Result] Desilets J, Zakhari A, Chagnon M, Ekmekjian T, Nguyen DB, Smith JP, Mansour FW, Krishnamurthy S. Pharmacologic Interventions to Minimize Fluid Absorption at the Time of Hysteroscopy: A Systematic Review and Meta-analysis. Obstet Gynecol. 2023 Feb 1;141(2):285-298. doi: 10.1097/AOG.0000000000005051. Epub 2023 Jan 4. PMID 36649319
- [Result] Welch K, Ek R, Stromme M. Comparative drug release measurements in limited amounts of liquid: a suppository formulation study. Curr Drug Deliv. 2006 Jul;3(3):299-306. doi: 10.2174/156720106777731109. PMID 16848731
- [Result] Bianchi M, Capurso L. Effects of guar gum, ispaghula and microcrystalline cellulose on abdominal symptoms, gastric emptying, orocaecal transit time and gas production in healthy volunteers. Dig Liver Dis. 2002 Sep;34 Suppl 2:S129-33. doi: 10.1016/s1590-8658(02)80180-3. PMID 12408456
- [Result] Vilos GA, Vilos AG, Abu-Rafea B, Ternamian A, Laberge P, Munro MG. Good practice with fluid management in operative hysteroscopy. Int J Gynaecol Obstet. 2025 Jan;168(1):118-125. doi: 10.1002/ijgo.15860. Epub 2024 Aug 22. PMID 39171580
- See also: Safety of Misoprostol — https://www.fda.gov/drugs/postmarket-drug-safety-information-patients-and-providers/misoprostol-marketed-cytotec-information
- See also: Microcrystalline Cellulose — https://www.researchgate.net/publication/334717784_Microcrystalline_Cellulose_as_Pharmaceutical_Excipient